CLINICAL TRIAL: NCT02151214
Title: Prospective, Multicenter, Randomized Controlled Study Evaluating the Efficacy of Parenteral Nutrition on the Quality of Life and Overall Survival in Patients in the Palliative Phase of Cancer.
Brief Title: Efficacy of Parenteral Nutrition in Patients at the Palliative Phase of Cancer.
Acronym: ALIM-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Institut Curie (Other); Institut de Cancérologie de Lorraine (Other); Centre Paul Strauss (Other); Institut Jean-Godinot (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Institut Paoli-Calmettes (Other); Centre Leon Berard (Other); Henri Mondor University Hospital (Other); Centre Oscar Lambret (Other); Centre Georges Francois Leclerc (Other); Centre Francois Baclesse (Other); Hôpital de la Timone (MARSEILLE) (Unknown)
Responsible Party: Principal Investigator, Régis AUBRY, Pr, Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ALIM-K
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Nutrition Aspect of Cancer; End Stage Cancer
Keywords: Palliative Phase of Cancer; Quality of life; Parenteral nutrition; Undernutrition
MeSH Terms: conditions — Hyperphagia; Malnutrition | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenteral nutrition (Experimental): Parenteral nutrition will be administered to the patients
  Interventions: Other: Parenteral nutrition
- Normal per os nutrition (No Intervention): The patients will eat orally

INTERVENTIONS:
Other: Parenteral nutrition — Administration of standard intravenous nutritional products. The products are commonly used in the department where the research is conducted
  Arms: Parenteral nutrition

SUMMARY:
In malnourished patients in the palliative phase of cancer, the question is raised of the relevance of implementing artificial nutritional assistance instead of oral feeding when this is possible.

Medical prescription and implementation of artificial nutrition at this stage of the illness seem less governed by data acquired by science than by subjective reasons (related to beliefs, to a cultural or religious tradition, to the symbolic role of eating, to the deeply ingrained fear of dying of hunger, to a portrayal of care, etc.) while interacting with teams, the patient and his family and relatives.

And yet, the benefits/risk balance and the effect on quality of life of parenteral nutrition in a palliative situation for patients presenting with a normal alimentary tract is poorly understood. The discomfort and risks of central venous or nasogastric artificial nutrition require that the benefits of artificial nutrition be proven. The nature of these benefits relate first and foremost to the quality of life experienced by the patient in such a context. Only a controlled randomized study may lead to an optimal palliative nutritional management of undernutrition to be determined, and to inform the patient and his/her relatives clearly in order for them to express their preferences.

We hypothesize that abstaining from artificial parenteral central venous nutrition and associated hydration for nutritional purposes improves quality of life without significant loss of survival compared to implementing artificial nutrition, when considered, in the absence of any specific curative treatment in anorexic patients in the palliative phase of cancer.

To test this hypothesis, we propose to carry out a multicenter, prospective, controlled, randomized study in order to evaluate the efficacy of implementing parenteral nutrition compared to abstaining from doing so on the quality of life of undernourished patients in the palliative phase of cancer. The effect on overall survival and the nutritional parameters will be evaluated.

The ALIM K trial will be carried out in 13 centres specializing in supportive and onco-hematology care .

ELIGIBILITY:
Inclusion criteria are:

* adult patients (aged >18 years) suffering from cancer at the palliative stage, i.e. patients in whom the main aim of treatment is to limit pain and discomfort
* curative treatment has either been discontinued, or may still be ongoing but with little expected benefit in terms of overall survival
* patients must already have a functional central venous catheter in place
* present malnutrition defined as a body mass index (BMI) <18.5 kg/m² in patients aged <70 years or <21 kg/m² in patients aged ≥70 years; or weight loss of 2% in 1 week, 5% in 1 month, or 10% in 6 months
* patients must have a functional digestive tract
* patients able to express themselves easily in French and answer questionnaires

Exclusion Criteria:

* Any condition that prevents orally feeding (especially patients with cancer of the upper aero-digestive tract, esophagus, obstructive stomach)
* Peritoneal carcinomatosis if it causes symptoms of sub-occlusion or bowel obstruction
* Non functional digestive tract (bowel obstruction, tumor compression)
* Patients with haematological cancers undergoing bonemarrow transplant,
* Life expectancy is less than 1 month
* Any contraindications to the parenteral nutrition prescription
* Parenteral nutrition that is ongoing or dating from less than one month;
* Presence of gastrostomy or jejunostomy;
* Persisting sensation of hunger in aphagic patients
* Patients participating in another ongoing clinical trial Adult
* Patients under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
QLQ-C15-Pal to assess Quality of Life through the physical functioning, Global Health Status and fatigue subscales | Time until definitive quality of life score deterioration
  The EORTC -The European Organisation for Research and Treatment of Cancer QLQ-C15-Pal - Quality of Life Questionnaire Core 15 Palliative is used.
  Physical functioning, global health status and fatigue are compared between the 2 groups.

SECONDARY OUTCOMES:
QUAL-E Measuring Quality of Life at the end of Life | Time until definitive quality of life score deterioration
  Questionaire for patients who believe they are nearing the end of life and comparison between the 2 groups.
Overall survival | Time from randomization to death
  Comparison of overall survival between the 2 groups
Other (non-primary-end point) domains of the QLQ-C15-PAL questionnaire (pain, emotional function, nausea/vomiting, appetite, dyspnea, constipation, and sleep) | Time until definitive quality of life score deterioration
  Comparison of other domains of the QLQ-C15-PAL questionnaire between the 2 groups.
Body weight | Time until definitive quality of life score deterioration
  Body weight will be compared between the 2 groups .
Body Mass Index | Time until definitive quality of life score deterioration
  Body Mass Index will be compared between the 2 groups .

CONTACTS AND LOCATIONS:
Overall Officials: Regis Aubry, Prof., Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (13):
- France (13):
  - Palliative Care Unit - CHU Jean Minjoz, Besançon
  - Centre François Baclesse, Caen
  - Centre hospitalier Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli calmettes, Marseille
  - Hopital de la Timone, Marseille
  - Institut Curie, Paris
  - Insitut Jean Godinot, Reims
  - Centre Paul Strauss, Strasbourg
  - Centre de cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Pazart L, Cretin E, Grodard G, Cornet C, Mathieu-Nicot F, Bonnetain F, Mercier M, Cuynet P, Bouleuc C, Aubry R; ALIM-K study investigational group. Parenteral nutrition at the palliative phase of advanced cancer: the ALIM-K study protocol for a randomized controlled trial. Trials. 2014 Sep 24;15:370. doi: 10.1186/1745-6215-15-370. PMID 25248371
- [Derived] Bouleuc C, Garabige V, Grodard G, Anota A, Aubry R, Marchal T. Impact of parenteral nutrition on oral intake and eating pleasure in advanced cancer patients: A sub-analysis of a multicenter randomized controlled trial. Clin Nutr ESPEN. 2026 Jan 12;72:102905. doi: 10.1016/j.clnesp.2025.102905. Online ahead of print. PMID 41534624